CLINICAL TRIAL: NCT02679716
Title: Hemodynamic Computer-assisted Reconstruction of Pathological Changes at the Origin of the Ophthalmic Artery in Patients With Retinal Artery Occlusion
Brief Title: Reconstruction of Pathological Changes of the Ophthalmic Artery in Patients With Retinal Artery Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RAO
Record Dates: First submitted 2016-02-07; First posted 2016-02-10 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Retinal Artery Occlusion
MeSH Terms: conditions — Retinal Artery Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study group (Other): MRI of the cerebral arteries ist performed
  Interventions: Other: MRI of the cerebral arteries

INTERVENTIONS:
Other: MRI of the cerebral arteries — MRI of the cerebral arteries is performed

SUMMARY:
Retinal artery occlusions (RAO) cause deterioration in visual acuity and visual fields. In computational fluid dynamics (CFD) studies [1] 10% of ascending emboli caused RAO, the residual 90% embolized into the cerebral arteries. As only 20% of patients with RAO had a history of stroke, there is a discrepancy between CFD-studies and clinical observations. Mead et al. [2] postulated small emboli being washed into the cerebral arteries without causing clinical symptoms of stroke, whereas similar emboli being washed into the ophthalmic artery would cause RAO.

There is a discrepancy between CFD-study results and clinical observations in RAO patients, indicating that there could be a high number of RAO-patients having had cerebral ischemies without symptoms of stroke (as postulated by Mead et al.[2]).

Purpose of the present study is to evaluate hemodynamic pathological changes at the ophthalmic artery origin in patients with RAO detected with an already existing CFD-model

DETAILED DESCRIPTION:
Retinal artery occlusions (RAO) cause deterioration in visual acuity and visual fields. Emboli from plaques of the carotid artery, aortic arch or vegetations of the cardiac valves are the main reasons for RAO. In computational fluid dynamics (CFD) studies [1] 10% of ascending emboli caused RAO, the residual 90% embolized into the cerebral arteries. As only 20% of patients with RAO had a history of stroke, there is a discrepancy between CFD-studies and clinical observations. Mead et al. [2] postulated small emboli being washed into the cerebral arteries without causing clinical symptoms of stroke, whereas similar emboli being washed into the ophthalmic artery would cause RAO. Hayreh et al. [3] reported plaques of the carotid artery to be the main reason for emboli causing RAO.

There is a discrepancy between CFD-study results and clinical observations in RAO patients, indicating that there could be a high number of RAO-patients having had cerebral ischemies without symptoms of stroke (as postulated by Mead et al.[2]). A recently published report showed ischemic cerebral lesions in 38% of patients with RAO without neurological symptoms [4]. The fact, that the 3-year risk of patients with RAO to develop stroke is doubled [5], underlines further associations between RAO and stroke.

Purpose of the present study is to evaluate hemodynamic pathological changes at the ophthalmic artery origin in patients with RAO detected with an already existing CFD-model

References (detailed references are provided in the reference section) :

[1] Leisser et al., [2] Mead et al., [3] Hayreh et al., [4] Lee et al., [5] Chang et al.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed RAO
* Older than 21 years
* Informed consent

Exclusion Criteria:

* Women in reproductive age

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Pathological changes in subjects with retinal artery occlusions | one hour
  assessed by magnetic resonance imaging

SECONDARY OUTCOMES:
number of patients with preexisting stroke | one hour
  assessed by medical history and magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Leisser, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery; Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery; Nino Hirnschall, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (2):
- Austria (2):
  - Vienna Institute for Research in Ocular Surgery, Vienna
  - Hanusch-Krankenhaus, Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leisser C, Kaufmann TA, Feltgen N, Schumacher M, Schmoor C, Meckel S. Distribution of internal carotid artery plaque locations among patients with central retinal artery occlusion in the Eagle study population. Graefes Arch Clin Exp Ophthalmol. 2015 Aug;253(8):1227-30. doi: 10.1007/s00417-014-2804-2. Epub 2014 Dec 13. PMID 25500982
- [Background] Mead GE, Lewis SC, Wardlaw JM, Dennis MS. Comparison of risk factors in patients with transient and prolonged eye and brain ischemic syndromes. Stroke. 2002 Oct;33(10):2383-90. doi: 10.1161/01.str.0000029827.93497.97. PMID 12364725
- [Background] Hayreh SS, Podhajsky PA, Zimmerman MB. Retinal artery occlusion: associated systemic and ophthalmic abnormalities. Ophthalmology. 2009 Oct;116(10):1928-36. doi: 10.1016/j.ophtha.2009.03.006. Epub 2009 Jul 3. PMID 19577305
- [Background] Lee J, Kim SW, Lee SC, Kwon OW, Kim YD, Byeon SH. Co-occurrence of acute retinal artery occlusion and acute ischemic stroke: diffusion-weighted magnetic resonance imaging study. Am J Ophthalmol. 2014 Jun;157(6):1231-8. doi: 10.1016/j.ajo.2014.01.033. Epub 2014 Feb 4. PMID 24503410
- [Background] Chang YS, Jan RL, Weng SF, Wang JJ, Chio CC, Wei FT, Chu CC. Retinal artery occlusion and the 3-year risk of stroke in Taiwan: a nationwide population-based study. Am J Ophthalmol. 2012 Oct;154(4):645-652.e1. doi: 10.1016/j.ajo.2012.03.046. Epub 2012 Jul 17. PMID 22809785